CLINICAL TRIAL: NCT03976648
Title: A Multicenter, Open-label Extension Study to Evaluate the Long-term Safety, Tolerability and Efficacy of Orally Administered GLPG1690 in Subjects With Systemic Sclerosis
Brief Title: A Clinical Study to Test Long Term Safety of GLPG1690 for Patients With Systemic Sclerosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The benefit-risk profile no longer supports continuing the studies
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GLPG1690-CL-206; 2019-001279-34 (EudraCT Number)
Record Dates: First submitted 2019-06-04; First posted 2019-06-06 (Actual); Results first posted 2022-03-15 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic | interventions — GLPG1690

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GLPG1690 600 mg (Experimental): Participants who received GLPG1690 600 milligrams (mg) in the GLPG1690-CL-204 (NCT03798366) study received GLPG1690 600 mg orally once daily up to 91 weeks.
  Interventions: Drug: GLPG1690
- Placebo (Experimental): Participants who received placebo matched to GLPG1690 in the GLPG1690-CL-204 (NCT03798366) study received GLPG1690 600 mg orally once daily up to 91 weeks.
  Interventions: Drug: GLPG1690

INTERVENTIONS:
Drug: GLPG1690 — film-coated tablets of GLPG1690 to be administered orally

SUMMARY:
This study was the extension of the double-blind study GLPG1690-CL-204 (NCT03798366). The main purpose of the study was to see how GLPG1690 was tolerated in participants with systemic sclerosis and whether there were any side effects in a long-term treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants who completed the 24-week treatment period of Study GLPG1690-CL-204 and who according to the investigator's judgment may benefit from long-term treatment with GLPG1690.

Exclusion Criteria:

* Any condition or circumstances that, in the opinion of the investigator, may make a participant unlikely or unable to complete the study or comply with study procedures and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-07-18 (Actual); Primary Completion 2021-04-13 (Actual); Study Completion 2021-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Galapagos Study Director, Study Director — Galapagos NV
Locations (14):
- United States (6):
  - Pacific Arthritis Care Center, Los Angeles, California
  - UCLA Rheumatology, Los Angeles, California
  - RASF Clinical Research Center, Boca Raton, Florida
  - University of Michigan, Ann Arbor, Michigan
  - Metroplex Clinical Research Center, Dallas, Texas
  - UT Physicians Center for Autoimmunity, Houston, Texas
- Belgium (2):
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
- Italy (2):
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Ospedale San Raffaele S.r.l. - PPDS, Milan
- Spain (2):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
- United Kingdom (2):
  - University Hospital Aintree, Liverpool
  - Royal Free Hospital, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Belgium, Italy, Spain, the United Kingdom, and the United States. The first participant was screened on 18 Jul 2019. The last study visit occurred on 13 Apr 2021. The treatment duration was planned for 104 weeks but the study was terminated at 91 weeks.
Pre-assignment Details: A total of 31 participants who completed 24-week double-blind treatment in the GLPG1690-CL-204 (NCT03798366) study were rolled over and randomized in this study.
Period: Overall Study
Arm/Group | GLPG1690 600 mg | Placebo
Started | 21 | 10
Completed | 0 | 0
Not Completed | 21 | 10
Not completed — Adverse Event | 0 | 2
Not completed — Study terminated by sponsor | 21 | 8

BASELINE CHARACTERISTICS:
Population: The open-label extension (OLE) full analysis set (FAS) was defined as all participants who had at least one intake of investigational product in the OLE study.
Groups:
- GLPG1690 600 mg: Participants who received GLPG1690 600 mg in the GLPG1690-CL-204 (NCT03798366) study received GLPG1690 600 mg orally once daily up to 91 weeks.
- Total: Total of all reporting groups
Arm/Group | GLPG1690 600 mg | Placebo | Total
Number analyzed (Participants) | 21 | 10 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (13.58) | 49.4 (18.57) | 50.1 (15.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 6 | 21
  Male | 6 | 4 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 20 | 10 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 21 | 9 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An adverse event (AE) was any untoward medical occurrence in a participant administered study drug and which did not necessarily have a causal relationship with study drug. A treatment-emergent adverse event (TEAE) is any AE with an onset date on or after the start of stud drug intake and no later than 30 days after last dose of study drug, or any worsening of any AE on or after the start of stud drug intake. A serious AE was defined as an AE that resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was medically significant. Safety analysis set consisted of all randomized participants who received at least 1 dose of investigational product.
Time Frame: Day 1 up to 91 weeks
Population: Participants in the OLE-FAS were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GLPG1690 600 mg | Placebo
Number analyzed (Participants) | 21 | 10
Participants
  TEAEs | 21 | 10
  Serious TEAEs | 6 | 3

ADVERSE EVENTS:
Time Frame: Day 1 up to 91 weeks
Description: Participants in the OLE-FAS were analyzed.
Arm/Group | GLPG1690 600 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/10
Serious Adverse Events (participants affected / at risk) | 6/21 | 3/10
Other Adverse Events (participants affected / at risk) | 21/21 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GLPG1690 600 mg (N=21) | Placebo (N=10)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Leukopenia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal prolapse (Gastrointestinal disorders) | 0 (0) | 1 (2)
Female genital tract fistula (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Thyroid mass (Endocrine disorders) | 1 (2) | 0 (0)
Colonic abscess (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (2) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GLPG1690 600 mg (N=21) | Placebo (N=10)
Hot flush (Vascular disorders) | 0 (0) | 1 (1)
Raynaud's phenomenon (Vascular disorders) | 3 (5) | 0 (0)
Discomfort (General disorders) | 0 (0) | 1 (1)
Nodule (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (3) | 0 (0)
Pyrexia (General disorders) | 1 (3) | 1 (1)
Peripheral swelling (General disorders) | 4 (5) | 1 (1)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1)
Breast fibrosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Weight increased (Investigations) | 2 (3) | 0 (0)
Bundle branch block left (Cardiac disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 4 (4) | 0 (0)
Bundle branch block right (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 2 (3) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 2 (3)
Headache (Nervous system disorders) | 6 (6) | 2 (3)
Altered visual depth perception (Eye disorders) | 0 (0) | 1 (1)
Blepharitis (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 8 (13) | 4 (7)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric antral vascular ectasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (3) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Digital pitting scar (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Scleroderma associated digital ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 6 (14) | 1 (4)
Skin lesion (Skin and subcutaneous tissue disorders) | 5 (6) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (7) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0)
Lactose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dyslipidaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0)
Conjunctivitis (Infections and infestations) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Infected skin ulcer (Infections and infestations) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 2 (2) | 1 (1)
Pharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Suspected COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 5 (7) | 1 (1)
Urinary tract infection (Infections and infestations) | 6 (11) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (6) | 1 (1)

LIMITATIONS AND CAVEATS:
The benefit-risk profile no longer supports continuing the studies. Therefore, the study was terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must review and approve any results of the study or abstracts for professional meetings prepared by the investigator(s). Published data must not compromise the objectives of the study. Data from individual study centers in multicenter studies must not be published separately.

DOCUMENTS (2):
  • Study Protocol (2020-01-08): https://cdn.clinicaltrials.gov/large-docs/48/NCT03976648/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-13): https://cdn.clinicaltrials.gov/large-docs/48/NCT03976648/SAP_001.pdf